CLINICAL TRIAL: NCT06698159
Title: Wide-Antral Pulmonary Vein Isolation in Patients Undergoing Atrial Fibrillation Ablation with a Single-shot Technique: the WIDER-PVI Trial
Brief Title: Wide-Antral Pulmonary Vein Isolation in Atrial Fibrillation Ablation with a Single-shot Technique (WIDER-PVI)
Acronym: WIDER-PVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Daniel Rodríguez Muñoz, Principal Investigator, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WIDER-PVI
Record Dates: First submitted 2024-11-05; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation (Paroxysmal)
Keywords: atrial fibrilation; cryoballoon; cryoablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: The distribution of patients to each arm will be in a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: The operators will not be blinded and will be aware of patient randomisation, which is necessary for the performance of the ablation procedure. The patient participant and the recurrence evaluation committee will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control strategy (Active Comparator): Pulmonary vein isolation by 28 mm balloon cryoablation
  Interventions: Device: Cryoablation with cryoballoon 28 mm
- Experimental strategy (Experimental): Pulmonary vein isolation by 31 mm balloon cryoablation
  Interventions: Device: Cryoablation with cryoballoon 31 mm

INTERVENTIONS:
Device: Cryoablation with cryoballoon 28 mm — Pulmonary vein isolation using 28 mm balloon cryoablation
  Arms: Control strategy
Device: Cryoablation with cryoballoon 31 mm — Pulmonary vein isolation using 31 mm balloon cryoablation
  Arms: Experimental strategy

SUMMARY:
The WIDER PVI study is a multicentre randomized clinical trial to compare the efficacy of antral versus extended antral PVI in patients with paroxysmal or persistent AF undergoing this procedure using a cryoablation balloon capable of 28 mm diameter (antral isolation) or 31 mm diameter (extended antral isolation) applications. The aim is to evaluate an objective of superiority of the extended antral isolation strategy versus antral isolation in the recurrence of atrial tachyarrhythmias at 1-year follow-up, both in episodes of >30 seconds duration and in overall arrhythmic load.

DETAILED DESCRIPTION:
Ablation has become a first-line therapy in the rhythm control strategy for atrial fibrillation (AF).

Pulmonary vein electrical isolation (PVI) is the cornerstone of ablation therapy, based on its efficacy profile, safety and lack of alternatives.

Single shot techniques have been increasingly used as the initial approach for PVI, employing cryoablation, i.e. release of cryoenergy into the endocardium via an inflatable catheter, to achieve isolation.

The most commonly used diameter in cryoablation is 28 mm. These generate antral isolation whose profile depends on the distance between veins. When the application is made with larger devices, as has been observed with the cryoballoon with an expandable diameter of 31 mm or ablation devices using pulsed electric fields, the isolation is also antral at the level of the carina, making the result of PVI more similar to that obtained when ablation is performed with a Wide Antral Circumferential Ablation (WACA) strategy using point-to-point radiofrequency (the gold standard for PVI).

The WIDER-PVI study aims to answer the question of whether single-shot ablation with a 31 mm diameter device is superior to conventional ablation with a 28 mm diameter device. The answer to this question is relevant in the context of the development of new, larger devices and concerns about the impact of larger ablation on atrial function.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Previous diagnosis of paroxysmal or persistent atrial fibrillation less than 2 years after diagnosis.
* Clinical indication to undergo a pulmonary vein isolation procedure using balloon cryoablation.

Exclusion Criteria:

* Severe left atrial dilatation (indexed volume >48 ml/m2 or area >40 cm2 or indexed diameter >3.0 cm/m2).
* Previous endocardial or surgical ablation of atrial fibrillation.
* Severe frailty (Clinical Frailty Scale score 7 or higher) or life expectancy less than 1 year.
* Inability to understand or give informed consent.
* Performance of other left atrial ablations in addition to pulmonary veins.
* Need to use another catheter in addition to the cryoablation catheter to complete pulmonary vein isolation.
* Contraindication to anticoagulation or intolerance to heparin.
* Presence of intra-atrial thrombus.
* Reversible cause of atrial fibrillation.
* Severe mitral or aortic valve disease.
* Congenital heart disease.
* Pregnancy or the prospect of pregnancy in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia | From enrollment to the end of follow up, assessed up to 12 months
  Presence of atrial fibrillation, atrial flutter, atrial tachycardia in which the atrial rate exceeds 180 beats per minute, lasting more than 30 seconds after the blanking period (8 weeks) and without pharmacological anti-arrhythmic treatment during 12 months of follow-up with continuous ECG monitoring (in patients with continuous implantable monitor) or combined (in patients without implantable monitor), by optical heart rate monitoring combined with programmed intermittent ECG and in response to detection of heart rate irregularity).
Arrhythmic load | From enrollment to the end of follow up, assessed up to 12 months
  Percentage of time the patient has atrial tachyarrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia in which the atrial rate exceeds 180 beats per minute) over the total monitored time.
Arrhythmic load | From 0 up to 60 minutes for every atrial tacharrhythmia detected in each patient
  Total duration of the longest episode of atrial tachyarrhythmia for each patient (cut off point: 60 minutes)

SECONDARY OUTCOMES:
Acute effectiveness | Every measure is assessed through procedure time, an average of 180 minutes
  * Percentage of veins in which complete occlusion (grade 4) is achieved pre-application
  * Percentage of veins requiring change to other than randomly assigned diameter
  * Percentage of patients in whom time to electrical isolation is visualised
  * Percentage of patients in whom pulmonary vein isolation is achieved at first application
  * Percentage of patients with termination of AF during applications, transitioning to sinus rhythm or to atrial tachycardia or flutter
Effectiveness in follow-up | Until the end of the study
  * Cardiovascular admissions
  * Visit to the emergency room for cardiovascular conditions
  * Death from any cause / death from cardiovascular cause
  * stroke/transient ischaemic attack
  * Percentage of patients requiring electrical or pharmacological cardioversion or new ablation for atrial tachyarrhythmia.
  * Percentage of patients with recurrence of AF after the blanking period and without pharmacological antiarrhythmic treatment.
  * Time to first recurrence of atrial tachyarrhythmia
  * Improvement in Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT) score from visit 0 (pre-ablation) to follow-up visit 12 months after ablation.
Safety | Until the end of the study
  * Major (death, complication requiring surgical or interventional treatment (vascular, coronary, cardiac, others) or prolongation of hospital stay >48 hours, or complication with chronic sequelae or requiring chronic treatment for its management) and minor adverse events
  * Intra-procedural complication rate
Acute effectiveness | Every measure is assessed through procedure time, an average of 180 minutes
  * Total procedure duration
  * Left atrial dwell time
  * Radiation exposure (fluoroscopy time and dose-area product)
  * Time to pulmonary vein electrical isolation

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (10):
  - IRCCS Neuromed Mediterranean Neurological Institute, Pozzilli, Isernia
  - Casa di cura Villa dei Fiori, Acerra, Napoli
  - Poliambulanza Institute Hospital Foundation, Brescia
  - Ospedale Santa Maria Goretti, Latina
  - Clinica San Michele, Maddaloni
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Pellegrini Hospital, Napoli
  - Department of Cardiac, Thoracic, Vascular Sciences and Public Health, University of Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, University "Cattolica del Sacro Cuore", Rome
  - S. Pietro Fatebenefratelli Hospital, Rome
- Spain (7):
  - HU Basurto, Bilbao
  - HU Virgen de las Nieves, Granada
  - HU Juan Ramón Jiménez, Huelva
  - Hospital Universitario 12 de Octubre, Madrid
  - HU Ramón y Cajal, Madrid
  - HU Virgen de la Victoria, Málaga
  - HU Virgen Macarena, Seville

REFERENCES:
- [Derived] Cobarro L, Negreira-Caamano M, Gomez-Burgueno L, Lopez-Alacid I, Ramos-Jimenez J, Marco Del Castillo A, Rajjoub Al-Mahdi EA, Borrego-Bernabe L, Estevez-Paniagua A, Boveda S, Delgado J, Salguero-Bodes R, Arribas-Ynsaurriaga F, Rodriguez-Munoz D. Wide-Antral pulmonary vein isolation in patients undergoing atrial fibrillation ablation with a Single-Shot technique: rationale and design of the WIDER-PVI trial. J Interv Card Electrophysiol. 2026 Jan;69(1):153-162. doi: 10.1007/s10840-025-02173-x. Epub 2025 Nov 6. PMID 41196540